CLINICAL TRIAL: NCT00093054
Title: Cranberry Juice and Urinary Tract Infections
Brief Title: Cranberry Juice for Treatment of Urinary Tract Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AT002086 (NIH)
Record Dates: First submitted 2004-09-30; First posted 2004-10-01 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Urinary Tract Infections
Keywords: Vaccinium macrocarpon
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cranberry juice
  Interventions: Drug: Cranberry juice
- 2 (Placebo Comparator): Placebo juice
  Interventions: Dietary Supplement: Placebo cranberry juice

INTERVENTIONS:
Drug: Cranberry juice — TID dosage for UTI treatment
  Arms: 1
Dietary Supplement: Placebo cranberry juice — TID placebo dosage to match active comparator
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether daily consumption of cranberry juice lessens the symptoms and prevents the recurrence of urinary tract infections (UTIs). This study will also determine whether drinking cranberry juice for 6 months selects for less virulent bacteria in the rectal, vaginal, and urethral areas.

DETAILED DESCRIPTION:
Participants in this study will be randomly assigned to consume either 8 ounces of cranberry juice or placebo juice twice a day for 6 months. Participants will have follow-up visits at 3 and 6 months, and whenever they experience a symptomatic episode. Urine, vaginal and rectal specimens will be taken at each visit to test for the presence of bacteria that cause urinary tract infections. Participants will complete a questionnaire at study entry, Day 3, Weeks 1 and 2, and monthly thereafter or whenever there is a recurrence of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Culture-confirmed urinary tract infection at study start

Exclusion Criteria:

* Other chronic disease
* Antibiotics within 48 hours prior to study start
* Hospitalization for any reason within 2 weeks prior to study start
* Stones in urinary tract
* Plans to leave Ann Arbor within 6 months after study start
* Allergy to cranberry or cranberry compounds
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Culture | per visit

CONTACTS AND LOCATIONS:
Overall Officials: Cibele T. Barbosa-Cesnik, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States